CLINICAL TRIAL: NCT00274040
Title: A Comparison of 18 μg of Tiotropium Inhalation Capsules and Atrovent Metered Dose Inhaler (2 Puffs of 20 μg, 4 Times Daily) in a Double-Blind, Double-Dummy, Efficacy and Safety Study in Adults With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Comparison of Tiotropium and Ipratropium in a Double-Blind, Double-dummy, Efficacy and Safety Study in Adults With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.244
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; Ipratropium

INTERVENTIONS:
Drug: Tiotropium
Drug: Ipratropium

SUMMARY:
Comparison of 18 mcg of Tiotropium Inhalation Capsules and ipratropiumMetered Dose Inhaler (2 puffs of 20 mcg, four times daily) in a Double-Blind, Double-dummy, Efficacy and Safety Study in Adults with Chronic Obstructive Pulmonary Disease (COPD).

The objective of this study is to compare the bronchodilator efficacy and safety of tiotropium inhalation capsules (18 mcg once daily) and ipratropium MDI (2 puffs of 20 mcg q.i.d.) in patients with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This is a 2-treatment, randomized, double-blind, parallel design trial in adult patient with COPD.

Each dose of tiotropium or placebo will consist of one capsule self administered from the HandiHaler device once daily during the treatment period (tiotropium or placebo). Each dose will be taken at the same time each morning between 08:00 a.m. and 10:00 a.m.

Each dose of ipratropium MDI or placebo MDI will consist of 2 puffs; patients will inhale 2 puffs four times daily. The first dose will be taken at the same time each morning between 08:00 a.m. and 10:00 a.m.; subsequent doses will be taken at lunch, at dinner and when going to bed.

Study Hypothesis:

The null hypothesis is that there is no difference in mean response between tiotropium and ipratropium.

The alternative hypothesis is that there is a difference in mean response between tiotropium and ipratropium.

Comparison(s):

This is a multi-center, randomized, double-blind, double-dummy, parallel group trial to compare the bronchodilator efficacy and safety of Tiotropium (18 mcg once a day) and ipratropium Metered Dose Inhaler (2 puffs of 18 mcg four times a day).

ELIGIBILITY:
Inclusion Criteria

1. All patients must have a diagnosis of chronic obstructive pulmonary disease according to the following criteria:

   Patients must have relatively stable airway obstruction with an FEV1 >= 65% of predicted normal and FEV1 70% of FVC. "Predicted normal values will be based on formulas as supplied by the individual study sites."
2. Male or female patients 40 years of age or older.
3. Patients must have a smoking history of more than 10 pack-years. A pack-year is defined as the equivalent of smoking one pack of cigarettes per day for a year.
4. Patients must be able to perform pulmonary function tests as required in the protocol.
5. Patients must be able to inhale medication from the HandiHaler device and should have a good technique of inhaling aerosol administered from an MDI.
6. All patients must sign an Informed Consent Form prior to participation in the trial i.e., prior to pre-study washout of their usual pulmonary medications

Exclusion Criteria

1. Patients with significant diseases other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
2. Patients with clinically significant abnormal baseline hematology, blood chemistry or urinalysis, if the abnormality defines a disease listed as an exclusion criterion will be excluded.
3. All patients with a SGOT and SGPT twice the normal range, bilirubin 150% or creatinine 125% of the normal range will be excluded regardless of the clinical condition. Repeat laboratory evaluation will not be conducted in these subjects.
4. Patients with a recent history (i.e. one year or less) of myocardial infarction.
5. Patients with a recent history (i.e. three years or less) of heart failure or patients with any cardiac arrhythmia requiring drug therapy.
6. Patients with regular use of daytime oxygen therapy.
7. Patients with known active tuberculosis.
8. Patients with a history of cancer within the last five years. Patients with treated basal cell carcinoma are allowed.
9. Patients with a history of life-threatening pulmonary obstruction, or a history of cystic fibrosis or bronchiectasis.
10. Patients who have undergone pulmonary resection or a thoracotomy for any reason.
11. Patients with an upper respiratory tract infection in the past 6 weeks prior to the Screening Visit (=Visit 1) or during the baseline period of 2-weeks (run-in period).
12. Patients with known hypersensitivity to anticholinergic drugs, lactose or any other component of the inhalation capsule delivery system or the MDI
13. Patients with known symptomatic prostatic hypertrophy or bladder neck obstruction.
14. Patients with known narrow-angle glaucoma.
15. Patients who are being treated with cromolyn sodium or nedocromil sodium.
16. Patients who are being treated with antihistamines.
17. Patients using oral corticosteroid medication at unstable (i.e. less than 6 weeks on a stable dose) or at a dose in excess of the equivalent 10 mg of prednisone per day or 20 mg every other day.
18. Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (e.g. oral contraceptives, intrauterine devices, or diaphragm).
19. Patients with a history of asthma, allergic rhinitis or atopy or who have a blood total eosinophil count 400>= per mcl (males) or 320>= per mcl (females). A repeat eosinophil count will not be conducted in these patients.
20. Patients with a history and/or active alcohol or drug abuse.
21. Patients who have taken an investigational drug one month or six half-lives (whichever is greater) prior to the Screening Visit (=Visit 1).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141
Dates: Start 2002-07; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Trough FEV1 response: change from baseline FEV1 (visit 2) to visit 4 trough FEV1 | 4 weeks

SECONDARY OUTCOMES:
FEV1 (AUC0-3) response (change from baseline) for the 3 hours post drug administration | 4 weeks
Trough FVC response | 4 weeks
FVC (AUC0-3) response (as defined for FEV1) | 4 weeks
Patient questionnaire | 4 weeks
Daily PEFR | 4 weeks
Amount of rescue medication | 4 weeks
All adverse events | 4 weeks
Vital signs (pulse rate and blood pressure) | 4 weeks
Number of patients with abnormalities in routine blood chemistry, haematology and urinanalysis | 4 weeks
Changes from baseline in 12-lead electrocardiogram (ECG) | 4 weeks
Physical examination | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Korea Ltd.
Locations (18):
- South Korea (18):
  - Chungnam National University Hospital, Daejeon
  - Jeonbuk National University Hospital, Jeonju
  - Jeonnam National University Hospital, Kwangju
  - Pusan University Hospital, Pusan
  - Chung-ang University Hospital, Seoul
  - Hanyang University Hosital, Seoul
  - Kangnam St. Mary's Hospital, Seoul
  - Korea University Hospital, Seoul
  - Kyoungbuk National University Hospital, Seoul
  - Kyunghee University Hospital, Seoul
  - National Medical Center, Seoul
  - Samsung Seoul Hospital, Seoul
  - Seoul Asan Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Shinchon Severence Hosp (Yonsei University Hosp), Seoul
  - St. Paul's Hospital, Dept. of Respiratory, Seoul
  - Youngdong Sevarence Hospital (Yonsei University Hospital), Seoul
  - Wonju Christian Hospital (Yonsei University Hosp), Wŏnju